CLINICAL TRIAL: NCT06129695
Title: Evaluation of Computer Guided Placement of Zygomatic Implants for Reconstruction of Atrophic Maxilla Utilizing Two Different Approaches: A Randomized Controlled Clinical Trial
Brief Title: Computer Guided Placement of Zygomatic Implants in Two Different Approaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdulrahman Adnan Aldakka, Master's degree candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A.A.D
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Atrophic Maxilla; Zygomatic Implants
Keywords: Zygoamtic implants, Dental implants, Atrophic maxilla, Intra sinus, Extra sinus and Full mouth rehabilitation
MeSH Terms: conditions — Atrophic Maxilla

STUDY DESIGN:
Intervention Model Description: 1. Randomized Controlled Clinical Trial.
  2. Parallel group study.
  3. Allocation Ratio 1:1.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each patient will be given a code by the researcher and the observers will be blind to which group this case belong. Patients, radiographic outcome assessor and statistician will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer guided intra sinus approach for Zygomatic implant placement. (Experimental): After reflection of mucoperiosteal flap then the non-working tip of the coarse diamond bur will be inserted till the initial marking point and further preparation of osteotomy site will be performed along the lateral wall of maxillary sinus then sinus membrane will be reflected gently to get easily access for 3.5 mm drill or 4-4.5 mm diameter Zygomatic implant. The surgical stent will be inserted inside the patient's mouth; it will be adapted and held in place by the anchoring screws to Zygoma and osteotomy will progressively widened by using standard 2.9 mm diameter drill and 3.5 mm twist diameter drill.
  Depth indicator will be used to determine the length of Zygomatic implant. Zygomatic implant will be placed.
  The platform of Zygomatic implant will be emerged over and close to the top of the crest of the residual alveolar ridge near to first molar region. Closure will done with 3-0 silk suture.
  Interventions: Procedure: Zygomatic implants
- Computer guided extra sinus approach for Zygomatic implant placement. (Active Comparator): After adequate exposure of surgical The surgical stent will inserted inside the patient's mouth; it will adapted and held in place by the anchoring screws to Zygoma and osteotomy will progressively widened by using standard 2.9 mm diameter drill and 3.5 mm twist diameter drill.
  Depth indicator will be used to determine the length of Zygomatic implant. Zygomatic implant that will placed.
  The platform of Zygomatic implant will be emerged over and close to the top of the crest of the residual alveolar ridge near to first molar region. Closure will done with 3-0 silk suture.
  Interventions: Procedure: Zygomatic implants

INTERVENTIONS:
Procedure: Zygomatic implants — the ideal way to support implant-based restorative procedures for full and partially edentulous patients who are missing bone in the upper posterior maxilla.

SUMMARY:
Evaluation of computer guided placement of Zygomatic implants utilizing intra sinus versus extra sinus surgical approach for the reconstruction of atrophic maxilla. The expected benefit from the current study is to select the most suitable approach for Zygomatic implant placement with the least postoperative complications

DETAILED DESCRIPTION:
During the last ten years, there has been an increase in the number of edentulous patients looking for and seeking out rehabilitation. Formerly, individuals with edentulous maxilla and mandibles were rehabilitated with removable complete dentures, but it was associated with poor patients' satisfaction.

Alveolar bone atrophy results from loss of bony support due to the physiological process that naturally takes place after tooth loss, especially in the upper arch. Due to its shape and structure, the maxilla is an extremely challenging arch to reconstruct with dental implants.

Oral and Maxillofacial surgeons began utilizing alternative methods to replace missing teeth with osseointegrated dental implants in atrophic maxilla. As a result, different methods were developed for handling of this issue, including tilted implants, sinus elevation, the use of Pterygoid implants, the use of short implants and Zygomatic implants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with severely atrophic edentulous upper arch (Cawood class IV, V, VI) that could not be restored by other type of treatment
2. Patients who had at least 8-12 mm vertical bone height in anterior maxilla to allow installation of 2 conventional implants.
3. Lacking posterior maxillary bone support due to significant sinus pneumatistion
4. Good systemic health (ASA score I-II)
5. Highly motivated patients.

Exclusion Criteria:

1. Patient not willing to give his/her informed consent.
2. Patients with systemic disease that did not permit the surgical procedure (including general anaesthesia).
3. Patients with uncontrolled diabetes or under bisphosphonate therapy.
4. Heavy smoker.(> 20 cigarettes daily)
5. Patient with psychiatric problems, severe bruxism or other parafunctional habits.
6. Acute sinusitis.
7. Malignancy or pathology in Maxilla or Zygoma.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2024-03-04 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Pain by Visual Analogue Scale (VAS) | operation day and first week
  1-10

SECONDARY OUTCOMES:
Crestal bone loss around zygomatic implants | after 6 months
  To measure the crestal bone loss around Zygomatic implant by CBCT.
Post operative complications | 1st week , first month , third month and sixth month
  Assessment of the incidence of the postoperative complications in the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Background] Ishak MI, Abdul Kadir MR, Sulaiman E, Abu Kasim NH. Finite element analysis of different surgical approaches in various occlusal loading locations for zygomatic implant placement for the treatment of atrophic maxillae. Int J Oral Maxillofac Surg. 2012 Sep;41(9):1077-89. doi: 10.1016/j.ijom.2012.04.010. Epub 2012 May 9. PMID 22575179
- [Background] Davo R, Malevez C, Rojas J. Immediate function in the atrophic maxilla using zygoma implants: a preliminary study. J Prosthet Dent. 2007 Jun;97(6 Suppl):S44-51. doi: 10.1016/S0022-3913(07)60007-9. PMID 17618933
- [Background] Jain DK, Pal US, Mohammad S, Mehrotra D, Katrolia R, Shandilya S, Yadav L, Tiwari AK. Comparative evaluation of extrasinus versus intrasinus approach for zygomatic implant placement. J Oral Biol Craniofac Res. 2022 Nov-Dec;12(6):863-872. doi: 10.1016/j.jobcr.2022.08.030. Epub 2022 Sep 10. PMID 36212616
- See also: Related Info — https://dialnet.unirioja.es/descarga/articulo/8822797.pdf